CLINICAL TRIAL: NCT05879146
Title: Evaluation of the Response and Non-response of Nirogacestat in Desmoid Tumors- Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0610; NCI-2023-04177 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nirogacestat (Experimental): Participants will take nirogacestat by mouth every day of each 28-day study cycle. Based on when you enroll in this study, you will take nirogacestat either 1 time a day at about the same time each day OR 2 times a day, about 12 hours apart.
  Interventions: Drug: Nirogacestat

INTERVENTIONS:
Drug: Nirogacestat — Given by PO

SUMMARY:
To learn about the safety and effects of an investigational drug called nirogacestat when given to participants with a desmoid tumor/aggressive fibromatosis

DETAILED DESCRIPTION:
Primary Objectives:

• To identify biomarkers associated with response and non-response to nirogacestat in participants with desmoid tumors (DT).

Secondary Objectives:

* To assess the 12-month progression-free survival (PFS of participants with DT who receive nirogacestat at 150 mg or 100 mg BID.
* To assess MRI volumetric and functional parameters associated with response and non-response to nirogacestat in participants with DT.
* To evaluate the histopathological changes in DT biopsy specimens.
* To evaluate the safety and tolerability of nirogacestat in participants with DT.

Exploratory Objectives:

* To assess clinical benefit and tumor response by additional MRI-based measurements including MRI-modified Choi criteria and WHO.
* To evaluate MRI parameters such as intensity histogram analysis from T2-weighted image (T2-WI), short inversion time inversion-recovery (T2-STIR), diffusion-weighted imaging (DWI) with apparent diffusion coefficient (ADC) mapping, post-contrast Water Dixon, perfusion-weighted imaging, and susceptibility-weighted imaging (SWI) with contrast and correlate with therapeutic response and clinical outcome.
* To assess the dynamics and concordance of circulating tumor cells (CTCs) in the blood compartment and tumor burden during nirogacestat treatment.
* To identify cell-free DNA (cfDNA) biomarkers associated with response and non-response to nirogacestat in patients with DT.
* To understand the impact of dose on the incidence of ovarian dysfunction in women of childbearing potential (WOCBP).

ELIGIBILITY:
Inclusion Criteria:

This study will enroll approximately 40 participants diagnosed with DT. Participants must meet the following eligibility criteria to be enrolled:

1. Age ≥ 18 years. Individuals younger than 18 years old are excluded. More than 99% of the population evaluated at MDACC with a diagnosis of DT is older than 18. Sixty-three percent of the population with a diagnosis of DT evaluated at MDACC are 10 - 54 years old. The remaining 37 percent are older than 54 years old. Additionally, most of the robust data related to dosing or adverse event data currently available on the use of nirogacestat is in adults
2. Histologically documented DT with evidence of radiographic tumor progression (≥ 10% or absolute increase in dimensions of ≥ 10 mm in maximal diameter) in unidimensional measurement within the previous 18 months. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam

   1. Recurrent or primary disease
   2. Symptomatic disease or impending morbidity (as defined by physician) and patient and physician agree treatment would be of benefit
3. Treatment naïve or progression on or after any prior therapy for DT. Participant must have discontinued prior therapy for at least 28 days or 5 half-lives of the drug, whichever is greater. All toxicities from prior therapy must be resolved to Grade ≤ 1 or clinical baseline. There is no limit on the number of previous systemic treatments received
4. Able to tolerate radiographic progression (up to 20% increase in tumor longest diameter) as determined by treating oncologist based on morbidity and tumor growth is not threatening vital structures
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Are appropriate for systemic therapy
7. Have accessible tumors for serial biopsies
8. Agree to provide new tumor tissue. Tumor tissue from the archival (tumor bank) may be used if the biopsy is performed after discontinuation of prior therapy and the participant must have discontinued prior therapy for at least 28 days or five half-lives of the drug, whichever is greater
9. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
10. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
11. Adequate organ and bone marrow function as defined by the following screening laboratory values:

    1. Absolute neutrophil count ≥ 1500 cells/μL;
    2. Platelets ≥ 100,000 μL;
    3. Hemoglobin ≥ 9 g/dL;
    4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%);
    5. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase)/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase) ≤ 2 × ULN; and
    6. If Creatinine > 1.5 x ULN then calculated creatinine clearance must be . 60 mL/min (using the Cockcroft-Gault formula).
12. Can swallow tablets and have no gastrointestinal conditions affecting absorption
13. Agree to the use of adequate contraception during the treatment period and for at least 4 months for men and women after the last dose of the study treatment (see Appendix 1 for more information)
14. Have the ability to understand and the willingness to sign a written informed consent document
15. English and non-English speaking patients
16. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this study
17. Participants with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification; to be eligible for this study, participants should be class 2B or better

Exclusion Criteria:

Participants are excluded from this study if any of the following criteria apply:

1. Unable to undergo serial biopsies
2. Participants with familial adenomatous polyposis
3. Unable to tolerate MRI or for whom MRI is contraindicated
4. Pregnant or breastfeeding women are excluded from this study. Based on findings in animal studies, oral administration of nirogacestat to pregnant rats during the period of organogenesis resulted in embryo-fetal toxicities at maternal exposures that were significantly lower than adult human exposures at the recommended dose of 150 mg twice daily. Nirogacestat should be avoided during pregnancy

   There is no data regarding the presence of nirogacestat or its metabolites in either human or animal milk or its effects on a breastfed child or on milk production. Because of the potential for serious adverse reactions in a breastfed child from nirogacestat, advise women not to breastfeed during treatment with nirogacestat.
5. Known hypersensitivity to nirogacestat or any of its excipients
6. Participants requiring the use of any excluded concomitant medications listed in Table 2 during the course of the study
7. Unable to comply with study-related procedures in the opinion of the investigator
8. Patients with cognitive impairment requiring a legally authorized representative for consent
9. Patients with uncontrolled intercurrent illness (Indicate clearly what type or extent)
10. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with positive viral load will be excluded
11. Patients with psychiatric illness/social situations that would limit compliance with study requirements
12. Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia
13. Patients who are receiving any other investigational agents
14. Patients with an additional malignancy and brain metastases. There is not enough evidence of the effects of nirogacestat in other malignancies at this time
15. Participant has experienced any of the following within 6 months of signing informed consent:

15.1 clinically significant cardiac disease (New York Heart Association Class III or IV); 15.2 myocardial infarction; 15.3 severe/unstable angina; 15.4 coronary/peripheral artery bypass graft; 15.5 symptomatic congestive heart failure; 15.6 cerebrovascular accident; 15.7 transient ischemic attack; or 15.8 symptomatic pulmonary embolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Keila Torres, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org